CLINICAL TRIAL: NCT05572346
Title: Use of a Digital App to Deliver Home-based Rehabilitative Interventions in Patients Affected by Respiratory Diseases: a Monocentric Observational Study
Brief Title: Digital App for Telerehabilitation in Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MedicAir Healthcare S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: RE-TEL
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Disease; Asthma; Long COVID; Chronic Obstructive Pulmonary Disease; Obesity; Lung Fibrosis; Bronchiectasis
Keywords: Respiratory Diseases; Telerehabilitation; Digital tools
MeSH Terms: conditions — Respiration Disorders; Asthma; Post-Acute COVID-19 Syndrome; Pulmonary Disease, Chronic Obstructive; Obesity; Pulmonary Fibrosis; Bronchiectasis; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Home-based telerehabilitation group: For each subject, the treatment will lasts 8 weeks. The intervention will include both endurance and resistance exercises as prescribed by the pneumologist at the time of the hospital discharge.
  The intervention will be delivered and monitored through a digital app with appropriate sensors.
  Interventions: Other: Home-based telerehabilitation program delivered through digital devices

INTERVENTIONS:
Other: Home-based telerehabilitation program delivered through digital devices — To evaluate the effects of digital home-based telerehabilitation program on functional and spirometric measures as well as on quality of life in patients with chronic respiratory disease

SUMMARY:
The purpose of this study is to evaluate the feasibility and the mid-term effects of a pulmonary rehabilitation intervention, delivered by digital App, on quality of life of patients affected by respiratory diseases. The App will include a monitored exercise training program based on most recent cardiopulmonary rehabilitation guidelines, including alerts, reminders and educational contents as well as chat and online visits with healthcare professionals to improve patient engagement.

DETAILED DESCRIPTION:
The center-based pulmonary rehabilitation (PR) intervention is considered the gold standard for functional recovery, secondary prevention, quality of life improvement and social as well as work reintegration in patients affected by respiratory diseases. Such kind of intervention, when delivered in all its fundamental components (clinical stabilization, functional assessment, physical and respiratory training, counseling, nutritional intervention and psychosocial support), is able to reduce global mortality and is recommended by the major international guidelines.

Despite the high level of recommendation, only a small fraction of patients after the acute hospital phase is currently initiated to PR programs for several reasons, including the limited number of specialized rehabilitation facilities.

This unmet need can cause a potential damage to patients' health (failure to reduce disability, higher risk of further pathological relapses) and generates an increase in social and healthcare costs, especially related to subsequent hospitalizations and loss of working capacity.

In order to fill the gap between PR need and demand, health systems are have to adopt not only organizational changes but also to implement innovative solutions based on new technologies. In particular, wearables and mobile health devices seem to be promising tools to deliver a sort of "light PR intervention" promoting healthier lifestyle, even in the long term.

Primary aim The primary objective of the study is to evaluate the feasibility and the medium-term effect on quality of life, measured by Visual Analogue Scale (VAS) contained in the EuroQoL 5D-5L questionnaire, of a digital home-based telerehabilitation program in patients with chronic obstructive pulmonary disease (COPD), asthma, bronchiectasis, pulmonary fibrosis, obesity and long COVID syndrome.

Secondary aims The secondary objectives are: to evaluate the impact of the intervention on functional capacity through the Six-Minute Walking test (6MWT); evaluate changes in dyspnea perception; evaluate the impact of the intervention on spirometric indices; evaluate adherence to the intervention delivered via digital app; evaluate usability, satisfaction, adverse events and exacerbations during the intervention delivered through the digital app.

Study design Monocentric, before-after study Assessment a baseline (T0) and after 8 weeks of intervention (T1)

Population 30 patients discharged from the Pulmonary Rehabilitation Unit of ICS Maugeri - IRCCS Lumezzane (Lumezzane - BS, Italy), affected by COPD, asthma, pulmonary fibrosis, bronchiectasis, obesity or long COVID syndrome.

Inclusion criteria Age ≥ 18 years old Diagnosis of COPD with Tiffenau index <70%, FEV1 <80%, asthma, bronchiectasis, pulmonary fibrosis, obesity (BMI > 30), long COVID syndrome Mini-mental status examination >22 Ability to perform a 6MWT with or without assistive devices Patients discharged from the Unit less than two weeks before the enrollment Written informed consent

Exclusion criteria Simultaneous participation to other research projects Simultaneous participation to other rehabilitation interventions High risk of heart failure and/or ventricular dysfunction High thrombotic risk Cardiac surgery within 3 months after the study enrollment High risk of arrhythmias Atrial fibrillation Moderate to severe valvulopathy Severe or not adequately controlled respiratory diseases Hemodynamic instability Anemia (Hb <10 g/dl) Pregnancy History of drugs abuse Total or partial inability to use digital devices Barriers to exercise training completion Full-day ventilotherapy

Materials and methods

At the hospital discharge (T0) a digital kit will be delivered in order to perform a home-based monitored telerehabilitation program. Using this kit, participants will undergo an 8-weeks exercise training and educational program to preserve the rehabilitative outcomes gained during hospital rehabilitation phase.

Every week participants will undergo a video-coaching session with a respiratory physiotherapist.

Primary endpoint Changes EuroQoL 5D-5L VAS score.

Secondary endpoint Change in COPD Assessment Test (CAT) and EuroQoL (VAS excluded) scores Variation of 6MWT performance at 8 weeks (T1) compared to T0 Variations of mean, maximal and at rest saturation during 6MWT at T1 compared to T0 Variations of mean, maximal and at rest heart rate as well as fatigue perception during 6MWT at T1 compared to T0 Change in Barthel Dyspnea and Medical Research Council (MRC) scores Variations of spirometric parameters: FVC, FEV1, Tiffeneau index, FEF75, FEF50, FEF25, FEF25-75 Adherence (number of sessions completed/number of sessions programmed ratio) Satisfaction and user experience assessment with Technology Acceptance Model (TAM) Assessment of adverse events and number of pathological relapses

Sample size Considering a Minimal Clinical Important Difference of 8 points at EuroQoL VAS, a standard deviation of 15 points, an alpha error of 5% and a power of 80%, the estimated sample size will be of 30 participants

Statistical analysis Data will be synthetized using descriptive statistics: quantitative variables will be summarized with means and standard deviations or medians and interquartile ranges, as appropriate; categorical variables will be expressed as absolute frequencies and percentages.

To assess outcomes changes following the 8-weeks intervention, parametric and non-parametric within group tests will be applied as appropriate.

Correlations between variables will be assessed using partial correlation analysis.

All the analyses will be conducted using SPSS 26 (IBM, Armonk, NY, USA).

Ethical and regulatory considerations This study will be conducted in accordance with the principles laid down by the 18th World Medical Assembly (Helsinki, 1964) and all applicable amendments laid down by the World Medical Assemblies, and the International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use (ICH) guidelines for Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD with Tiffenau index lower than 70%, FEV1 lower than 80%, asthma, bronchiectasis, pulmonary fibrosis, obesity (BMI higher than 30), long COVID syndrome;
* Mini-mental status examination higher than 22;
* Ability to perform a 6MWT with or without assistive devices;
* Patients discharged from the Pulmonary Rehabilitation Unit less than two weeks before the enrollment;
* Release of written informed consent

Exclusion Criteria:

* Simultaneous participation to other research projects;
* Simultaneous participation to other rehabilitation interventions;
* High risk of heart failure and/or ventricular dysfunction;
* High thrombotic risk;
* Cardiac surgery within 3 months after the study enrollment;
* High risk of arrhythmias;
* Atrial fibrillation
* Moderate to severe valvulopathy;
* Severe or not adequately controlled respiratory diseases;
* Hemodynamic instability;
* Anemia (Hb lower than 10 g/dl);
* Pregnancy;
* History of drugs abuse
* Total or partial inability to use digital devices
* Barriers to exercise training completion
* Full-day ventilotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients discharged from the Pulmonary Rehabilitation Unit of ICS Maugeri - IRCCS Lumezzane (Lumezzane - BS, Italia), affected by COPD, asthma, pulmonary fibrosis, bronchiectasis, obesity or long COVID syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Effects of home-based telerehabilitation intervention on self-perceived overall quality of life | 8 weeks
  Rating of EuroQoL 5D-5L Visual Analogue Scale (VAS) score changes: the EuroQoL 5D-5LVAS scale is a graduated line ranging from 0 (worse quality of life) to 100 (better quality of life). Longitudinal changes will be obtained subtracting baseline VAS to VAS at follow-up. A positive score means quality of life improvement, a negative score, a worsening of quality of life.

SECONDARY OUTCOMES:
Effects of home-based telerehabilitation intervention on quality of life | 8 weeks
  Assessment in COPD Assessment Test (CAT) and EuroQoL (VAS excluded) scores changes.
  Longitudinal changes will be obtained subtracting baseline score to follow-up score. A positive score means quality of life improvement, a negative score, a worsening in quality of life.
Effects of home-based telerehabilitation intervention on exercise tolerance | 8 weeks
  Assessment of six-minutes walking test (6MWT) changes: this is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. It is expressed in meters and ranges from 0 (worse performance) to infinity (better performance).
  Longitudinal changes will be obtained subtracting baseline distance to distance walked at follow-up. A positive score means walking improvement, a negative score, a worsening of walking ability.
Effects of home-based telerehabilitation intervention on heart rate | 8 weeks
  Assessment of heart rate changes (measured during 6MWT) at follow-up compared to baseline.
  Heart rate will be expressed as beats per minute
Effects of home-based telerehabilitation intervention on fatigue during exercise | 8 weeks
  Assessment of fatigue perception change during 6MWT at follow-up compared to baseline. Fatigue will be evaluated using Borg CR-10. A 10-points scale where 0 represents no effort and 10 maximal effort
Effects of home-based telerehabilitation intervention on dyspnea perception | 8 weeks
  Assessment of Barthel Dyspnea and Medical Research Council (MRC) scores changes at follow-up compared to baseline.
  Both scales measure the self-perceived dyspnea. Barthel ranges from 0 to 100, where lower scores represent worse clinical condition and 100 is the best condition.
  MRC ranges from 1 to 5 and lower scores represent a better clinical condition
Effects of home-based telerehabilitation intervention on forced vital capacity (FVC) | 8 weeks
  Assessment of FVC variations with spirometry measured in liters at follow up compared to baseline
Effects of home-based telerehabilitation intervention on forced expiratory volume in the first second (FEV1) | 8 weeks
  Assessment of FEV1 variations with spirometry measured in liters at follow up compared to baseline
Effects of home-based telerehabilitation intervention on Tiffeneau index | 8 weeks
  Assessment of Tiffeneau index variations measured with spirometry at follow up compared to baseline. The index is obtained by FEV1/FVC ratio and expressed as percentage.
Effects of home-based telerehabilitation intervention on forced expiratory flow (FEF) | 8 weeks
  Assessment of FEF index variations measured with spirometry at follow up compared to baseline. FEF will be assessed at 25% of FVC, 75% of FVC and FEF 25-75 (liters/seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Chiara G Beccaluva, MSc, Study Chair — MedicAir Italia S.r.l.; Michele Vitacca, MD, Principal Investigator — ICS Maugeri - IRCCS Lumezzane
Locations (1):
- ICS Maugeri - IRCCS Lumezzane, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No